CLINICAL TRIAL: NCT01091129
Title: Clinical Evaluation of the miraDry System in Subjects With Hyperhidrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Miramar Labs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-0004
Record Dates: First submitted 2010-03-19; First posted 2010-03-23 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Axillary Hyperhidrosis
Keywords: hyperhidrosis
MeSH Terms: conditions — Hyperhidrosis | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Treatment with the miraDry System in both axilla
  Interventions: Device: miraDry System (treatment with energy)

INTERVENTIONS:
Device: miraDry System (treatment with energy) — Treatment with microwave energy delivery device as specified by manufacturer's instructions
  Other Names: miraDry System

SUMMARY:
The purpose of this study is to determine whether treatment by the miraDry System can safely reduce the severity of axillary hyperhidrosis (excessive underarm sweating).

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years of age or older at the time of consent.
* Subject reports a quality-of-life rating of 3 or 4 on the Hyperhidrosis Disease Severity Scale.
* Subject has a baseline gravimetric measurement of spontaneous resting sweat production of at least 50mg/5min at room temperature in each axilla.
* Subject has primary focal axillary hyperhidrosis evidenced by at least two of the following:

  * Bilateral and relatively symmetric
  * Impairs daily activities
  * Frequency of at least one episode per week
  * Age of onset less than 25 years old
  * Positive family history
  * Cessation of focal sweating during sleep.
* In the opinion of the physician, treatment with the miraDry System is technically feasible and clinically indicated.
* Subject has provided written informed consent using a form that has been approved by the reviewing IRB/ethics committee.
* Subject is willing and able to comply with protocol requirements and all study visits.
* Female subjects of child-bearing potential must not be pregnant or lactating and must agree to not become pregnant during the course of the study.

Exclusion Criteria:

* Subject has secondary hyperhidrosis due to medications, infections, malignancy or endocrinopathy.
* Subject has hyperhidrosis on the trunk or chest.
* Subject has evidence of active infection.
* Prior endoscopic thoracic sympathectomy, liposuction or other surgery for axillary hyperhidrosis.
* Axillary injection of botulinum toxin within one year preceding the miraDry treatment.
* Oral anticholinergic medication use (e.g., Robinul) or cholomimetic medication use within the last 4 weeks or planned use during the study's follow up phase.
* Subject is a prisoner or under incarceration.
* Currently participating in or recently participated in another clinical trial (within the last 30 days).
* History of or current neurologic deficit in the treatment limb.
* Known resistance to or history of difficulty with local anesthesia (lidocaine with epinephrine).
* History of cancer with the exception of (1) successfully treated basal cell or squamous cell carcinoma of the skin or (2) subjects with a history of successfully treated cancer that have been disease-free for five years.
* Injury in the treatment area, shoulder or limb, which, in the opinion of the physician would render this subject an unacceptable candidate for DTS treatment (e.g., prior surgical repair, injury of the shoulder requiring physical therapy).
* Subject has a pacemaker, defibrillator or other electronic implant
* Subject requires supplemental oxygen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-02; Primary Completion 2011-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects that rate themselves as HDSS of 1 or 2 at the 30 day follow-up visit will be greater than 50% with a 95% confidence. | 30 days after final treatment session
Rate of serious adverse events | 12 months post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Chih-ho Hong, MD, Principal Investigator — Guildford Dermatology Specialists
Locations (2):
- Canada (2):
  - Guildford Dermatology Specialists, Surrey, British Columbia
  - Cosmedica, Victoria, British Columbia